CLINICAL TRIAL: NCT04429269
Title: A Comparative Study of Mammography and Ultrasound for Breast Cancer Screening and Early Diagnosis
Acronym: MUSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-MUSD
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Diagnosis; Breast Cancer Screening
Keywords: Mammography; ultrasound; breast cancer screening; early diagnosis
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy or specimen from volunteers or donors are planned to be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mammography and ultrasound: mammography and ultrasound screening
  Interventions: Diagnostic Test: mammography and ultrasound screening

INTERVENTIONS:
Diagnostic Test: mammography and ultrasound screening — Patients screened by both mammography and ultrasound.

SUMMARY:
Improving the early diagnosis of breast cancer can reduce mortality. With mammography as the main tool for screening early breast cancer, the characteristics of dense breast and young onset of disease in Chinese women lowers the efficiency. The aim of this prospective study was to compare which method, x-ray or ultrasound, is more appropriate for screening and early diagnosis of breast cancer in Chinese women.

DETAILED DESCRIPTION:
Breast cancer has become the most common malignancy in women. Improving the early diagnosis of breast cancer can reduce mortality. Mammography is recommended as the main tool for screening and early diagnosis of breast cancer in the guidelines of European and American countries. However, the characteristics of dense breast and young onset of disease in Chinese women make the screening and early diagnosis strategies of Western countries, which are mainly based on mammography, unsuitable for Chinese women. The aim of this prospective study was to compare which method, x-ray or ultrasound, is more appropriate for screening and early diagnosis of breast cancer in Chinese women.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, subjects 35-70 years old, asymptomatic, able to undergo ultrasound and x-ray

Exclusion Criteria:

* Localized breast erythema and ulceration, pregnancy, lactation, after previous breast implantation, already pathologically definite breast cancer patients

Ages: 35 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Chinese female subjects aged 35-70 years who were asymptomatic and able to undergo ultrasound and X-rays
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
screening yield | 3 years
  The sensitivity, specificity, positive predictive value, and negative predictive value of the screening methods.

SECONDARY OUTCOMES:
cost-effectiveness | 3 years
  The cost-effectiveness of each screening modality to detect one case of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Songjie Shen, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and PUMC, BJ, China
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual information of each participant of the trials is not shown in public, yet can be obtained upon reasonable requirements.

REFERENCES:
- [Derived] Wang Y, Li Y, Qu Y, Zhou Y, Sun Q, Shen S. Clinical and imaging characteristics of intraductal papillary neoplasms of the breast: a prospective trial. Discov Oncol. 2024 Dec 23;15(1):831. doi: 10.1007/s12672-024-01681-y. PMID 39715848
- [Derived] Wang Y, Li Y, Song Y, Chen C, Wang Z, Li L, Liu M, Liu G, Xu Y, Zhou Y, Sun Q, Shen S. Comparison of ultrasound and mammography for early diagnosis of breast cancer among Chinese women with suspected breast lesions: A prospective trial. Thorac Cancer. 2022 Nov;13(22):3145-3151. doi: 10.1111/1759-7714.14666. Epub 2022 Sep 30. PMID 36177910